CLINICAL TRIAL: NCT02576808
Title: Comparative Study of Efficacy and Adverse Effects of Ginger Extract and Loratadine for Treatment of Allergic Rhinitis Patients (Clinical Trial Phase II)
Brief Title: Study of Efficacy and Safety of Ginger Extract Compared With Loratadine for Treatment of Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thai Traditional Medical Knowledge Fund (Other Government)
Collaborators: Thammasat University (Other)
Responsible Party: Principal Investigator, Rodsarin Yamprasert, Faculty of Medicine Thammasat University, Thai Traditional Medical Knowledge Fund
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-EC-TM-4-077/57; TCTR20151001001 (Registry Identifier: Thai Clinical Trials Registry (TCTR))
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Rhinitis,Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — ginger extract; Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger extract (Experimental): Drug
  Interventions: Drug: Ginger extract
- Loratadine (Active Comparator): Drug
  Interventions: Drug: Loratadine

INTERVENTIONS:
Drug: Ginger extract — Ginger extract capsule at dose of 250 mg two times a day after meal daily for 42 days
  Arms: Ginger extract
Drug: Loratadine — Loratadine tablet at dose of 10 mg one times a day after morning meal daily for 42 days
  Other Names: Clarityne
  Arms: Loratadine

SUMMARY:
Efficacy and adverse effects of Ginger extract in treating allergic rhinitis patients compared with Loratadine.The double blind randomized controlled trial study was approved by the Human Research Ethics Committee of Thammasat University NO.1.

DETAILED DESCRIPTION:
The double blind randomized controlled trial study. Patients who meet the inclusion criteria and do not fall into any exclusion criteria will be randomly placed into the experimental group, who will receive ginger extract capsules, or the control group, who will receive loratadine for 42 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have moderate allergic rhinitis (itching and nasal obstruction, watery nasal discharge, sneezing and congestion )with a minimum total nasal symptom score 7 point
2. These patients do not have the respiratory disease such as tuberculosis, nasal polyps.
3. These patients do not have the history of disease: heart disease, kidney disease, liver disease, epilepsy, high blood pressure and severe asthma.
4. These patients are not pregnant or breastfeeding.
5. These patients have normal BMI and vital signs.

Exclusion Criteria:

1. Those who have taken anti-coagulant and anti-platelet aggregation medications.
2. Those who get serious side effects from Loratadine and ginger allergy.
3. Communication problems especially listening and interview.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Nasal symptom | 42days
  Nasal symptom from Total nasal symptom score

SECONDARY OUTCOMES:
Quality of Life | 42days
  Quality of Life from Rhinoconjunctivitis Quality of Life Questionnaire
Nasal patency | 42days
  Nasal patency from Acoustic rhinometry

CONTACTS AND LOCATIONS:
Overall Officials: Rodsarin Yamprasert, Principal Investigator — Faculty of Medicine Thammasat University (Rangsit Campus)
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yamprasert R, Chanvimalueng W, Mukkasombut N, Itharat A. Ginger extract versus Loratadine in the treatment of allergic rhinitis: a randomized controlled trial. BMC Complement Med Ther. 2020 Apr 20;20(1):119. doi: 10.1186/s12906-020-2875-z. PMID 32312261